CLINICAL TRIAL: NCT07319702
Title: Clinical Effects of Proprioceptive Neuromuscular Facilitation Combined With Spiral Muscle Chain Training in the Treatment of Children With Scoliosis
Brief Title: Proprioceptive Neuromuscular Facilitation Combined With Spiral Muscle Chain Training for Pediatric Scoliosis
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Nie danning (Other)
Responsible Party: Sponsor-Investigator, Nie danning, PhD Candidate, Nanjing Normal University
Organization: Nanjing Normal University (Other)
Allocation: Randomized | Model: Factorial | Masking: Double | Purpose: Treatment
Other Study IDs: NNU202410016
Record Dates: First submitted 2025-12-20; First posted 2026-01-06 (Actual); Last update posted 2026-01-06 (Actual); Status verified 2025-12

CONDITIONS: Adolescent Idiopathic Scoliosis (AIS)
Keywords: Adolescent Idiopathic Scoliosis; Proprioceptive Neuromuscular Facilitation; Spiral Muscle Chain Training; Exercise Therapy; Rehabilitation
MeSH Terms: interventions — Muscle Stretching Exercises; Therapeutics

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Proprioceptive Neuromuscular Facilitation (PNF) Therapy (Experimental): Participants receive proprioceptive neuromuscular facilitation (PNF) therapy as an exercise intervention for abnormal spinal curvature. Training is conducted 3 times per week (every other day) for 12 weeks. The PNF protocol includes resisted scapular-pelvic patterns, cervical flexion/extension, trunk chopping/lifting patterns, bilateral upper-limb patterns, and bridge exercises (per PNF schedule).
  Interventions: Behavioral: Proprioceptive Neuromuscular Facilitation (PNF) Therapy
- Spiral Muscle Chain (SPS) Training (Experimental): Participants receive spiral stabilizing muscle chain (SPS) training as an exercise intervention for abnormal spinal curvature. Training is conducted 3 times per week (every other day) for 12 weeks. The SPS program follows the SPS training schedule (Training 1A-6A, 7C-10C, and stretching component), with planned repetitions/sets and practice time as listed in the protocol schedule.
  Interventions: Behavioral: Spiral Muscle Chain (SPS) Training
- Combined Exercise Therapy (Experimental): Participants receive a combined program consisting of PNF therapy plus SPS spiral muscle chain training as an exercise intervention for abnormal spinal curvature. Training is conducted 3 times per week (every other day) for 12 weeks.
  Interventions: Behavioral: Combined Exercise Therapy

INTERVENTIONS:
Behavioral: Proprioceptive Neuromuscular Facilitation (PNF) Therapy — Proprioceptive neuromuscular facilitation (PNF) therapy is used as an exercise-based intervention to address abnormal spinal curvature in children with adolescent idiopathic scoliosis.
  The PNF program includes resisted scapular-pelvic patterns, cervical flexion and extension, trunk diagonal patterns (chopping and lifting), bilateral upper-limb diagonal patterns, and bridge exercises.
  Training sessions are supervised and conducted three times per week (every other day) for 12 weeks.
  Other Names: Proprioceptive Neuromuscular Facilitation
  Arms: Proprioceptive Neuromuscular Facilitation (PNF) Therapy
Behavioral: Spiral Muscle Chain (SPS) Training — Spiral muscle chain (SPS) training is applied as an exercise-based intervention aimed at improving spinal alignment, postural control, and neuromuscular coordination in children with adolescent idiopathic scoliosis.
  The SPS program consists of spiral stabilization exercises performed with elastic resistance, body positioning control, and stretching components according to a standardized training protocol.
  Training sessions are supervised and conducted three times per week (every other day) for 12 weeks.
  Other Names: Spiral Stabilization Training
  Arms: Spiral Muscle Chain (SPS) Training
Behavioral: Combined Exercise Therapy — The combined intervention integrates proprioceptive neuromuscular facilitation (PNF) therapy and spiral muscle chain (SPS) training as a comprehensive exercise program for children with adolescent idiopathic scoliosis.
  Participants perform both PNF and SPS exercise components within each training cycle to target spinal alignment, muscle endurance, and neuromuscular activation.
  Training sessions are supervised and conducted three times per week (every other day) for 12 weeks.
  Arms: Combined Exercise Therapy

SUMMARY:
The goal of this clinical trial is to evaluate the clinical effectiveness of proprioceptive neuromuscular facilitation (PNF) combined with spiral muscle chain (SPS) training in improving spinal function and posture in children with adolescent idiopathic scoliosis.

The main questions it aims to answer are:

Does PNF combined with SPS training improve trunk alignment and body balance parameters in children with mild adolescent idiopathic scoliosis?

Does the combined intervention improve spinal mobility and paraspinal muscle endurance compared with single-intervention approaches?

Does the combined intervention lead to favorable changes in surface electromyography (sEMG) indicators of trunk and paraspinal muscles?

Researchers will compare a PNF therapy group, an SPS training group, and a combined PNF + SPS group to assess differences in spinal alignment, muscle endurance, and neuromuscular activation outcomes.

Participants will:

Be assigned to one of three intervention groups: PNF therapy alone, SPS training alone, or combined PNF and SPS training

Participate in supervised exercise training sessions three times per week for 12 weeks

Undergo pre- and post-intervention assessments, including electronic spinal measurements and surface electromyography testing

ELIGIBILITY:
Inclusion Criteria:

- Age 13 to 18 years

Angle of trunk rotation (ATR) 5° ≤ ATR < 10°

No brace treatment and no history of spinal surgery

Able to complete PNF therapy and SPS training as required

Written informed consent obtained (participants and their parents/guardians)

Exclusion Criteria:

* Non-idiopathic scoliosis

Any exercise-related contraindications

History of spinal surgery

Any congenital deformity

Any trauma within the previous 6 months

Any accompanying neurological, rheumatological, or mental problems

Ages: 13 Years to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 189 (Actual)
Dates: Start 2024-03-05 (Actual); Primary Completion 2024-12-30 (Actual); Study Completion 2024-12-30 (Actual)

PRIMARY OUTCOMES:
Change in Trunk Tilt Angle (ATI) | Baseline and after 12 weeks of intervention
  Trunk tilt angle (Angle of Trunk Rotation, ATI) measured using an electronic spine assessment device to evaluate changes in spinal asymmetry and trunk alignment.
Change in Body Balance Parameters | Baseline and after 12 weeks of intervention
  Body balance parameters assessed by electronic spine measurement, including head lateral deviation, shoulder asymmetry, and pelvic tilt.
Change in Paraspinal Muscle Endurance | Baseline and after 12 weeks of intervention
  Paraspinal muscle endurance evaluated during the Biering-Sorensen test using surface electromyography-derived fatigue indicators.

SECONDARY OUTCOMES:
Change in Spinal Mobility | Baseline and after 12 weeks of intervention
  Spinal mobility assessed by electronic spine measurement, including lateral flexion, flexion-extension, and rotational range of motion.
Change in Surface Electromyography Parameters | Baseline and after 12 weeks of intervention
  Surface electromyography (sEMG) parameters including EMG amplitude, integrated EMG (iEMG), slope of median frequency (SlopeMF), and slope of mean power frequency (SlopeMPF) recorded from bilateral trapezius, erector spinae, and multifidus muscles.
Change in Trunk Muscle Activation Patterns | Baseline and after 12 weeks of intervention
  Trunk muscle activation patterns assessed during standardized functional tasks using surface electromyography.

CONTACTS AND LOCATIONS:
Locations (1):
- The Affiliated High School of Nanjing Normal University, Nanjing, Jiangsu, China

IPD SHARING:
Plan to Share IPD: No
Individual participant data (IPD) will not be shared because the study involves minors, and the data include sensitive health information related to spinal posture and neuromuscular function. According to the approved ethics protocol, strict measures are required to protect participants' privacy and confidentiality. Although all data are de-identified, sharing IPD may still pose a potential risk of re-identification. Therefore, IPD will not be made publicly available in order to ensure compliance with ethical requirements and data protection regulations.

REFERENCES:
- [Result] Xu Y, Feng M, Wu R, Wang Y, Yang Z, Wang Z, Kang Z, Xie L, Liu H. Effect of adding proprioceptive neuromuscular facilitation to conventional physiotherapy on scapular balance and shoulder proprioception in adolescents with idiopathic scoliosis: a randomised controlled trial protocol. BMJ Open. 2025 Nov 19;15(11):e106848. doi: 10.1136/bmjopen-2025-106848. PMID 41263915
- [Result] Nechvatal P, Hitrik T, Kendrova LD, Macej M. Comparison of the effect of the McKenzie method and spiral stabilization in patients with low back pain: A prospective, randomized clinical trial. J Back Musculoskelet Rehabil. 2022;35(3):641-647. doi: 10.3233/BMR-210055. PMID 34657873
- [Result] Maruyama T, Kitagawa T, Takeshita K, Mochizuki K, Nakamura K. Conservative treatment for adolescent idiopathic scoliosis: can it reduce the incidence of surgical treatment? Pediatr Rehabil. 2003 Jul-Dec;6(3-4):215-9. doi: 10.1080/13638490310001642748. PMID 14713588

DOCUMENTS (2):
  • Study Protocol (2024-03-01): https://cdn.clinicaltrials.gov/large-docs/02/NCT07319702/Prot_000.pdf
  • Informed Consent Form (2024-03-01): https://cdn.clinicaltrials.gov/large-docs/02/NCT07319702/ICF_001.pdf